CLINICAL TRIAL: NCT00646594
Title: A Two Stage Randomized, Open-Label, Parallel Group, Phase III, Multicenter, 7 Month Study to Assess the Efficacy & Safety of SYMBICORT pMDI Adminstered Either as Fixed or as an Adjustable Regimen Versus a Fixed Regimen of Advair in Subjects 12 Yrs of Age and Older With Asthma.
Brief Title: Atlantis Symbicort
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5896C00005
Record Dates: First submitted 2008-03-26; First posted 2008-03-28 (Estimated); Last update posted 2009-03-27 (Estimated); Status verified 2009-03

CONDITIONS: Asthma
Keywords: Asthma; inhaled cortocisteroids; Symbicort; budesonide/formoterol; Advair; fluticasone/salmeterol
MeSH Terms: conditions — Asthma | interventions — Budesonide; Formoterol Fumarate; Budesonide, Formoterol Fumarate Drug Combination; Fluticasone; Salmeterol Xinafoate; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): budesonide/formoterol
  Interventions: Drug: budesonide/formoterol (Symbicort)
- 2 (Active Comparator): fluticasone/salmeterol
  Interventions: Drug: fluticasone/salmeterol (Advair)

INTERVENTIONS:
Drug: budesonide/formoterol (Symbicort)
  Other Names: Symbicort
  Arms: 1
Drug: fluticasone/salmeterol (Advair)
  Other Names: Advair
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether Symbicort compared with Advair, will be more effective in controlling asthma in adults and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma
* Baseline lung function tests as determined by protocol
* Required and received treatment with inhaled corticosteroids within timeframe and doses specified in protocol

Exclusion Criteria:

* Has required treatment with any non-inhaled corticosteroid within previous 30 days, sensitivity to drugs specified in the protocol, or requires treatment with a beta-blockers
* Had cancer within previous 5 years or currently has any other significant disease or disorder as judged by the investigator

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2003-11; Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Asthma control assessed by asthma exacerbations | Continuosly throughout the treatment period

SECONDARY OUTCOMES:
Efficacy of Symbicort compared with Advair as assessed by use of rescue medication, asthma symptoms, lung function tests, quality of life reports, patient reported asthma control and patient satisfaction of Symbicort. | Daily and at 1, 3 and 6 months after start of treatmen
Use of medical resources and medication for the treatment of asthma. | Throughout the treatment period
Investigate safety profile of Symbicort compared to Advair | 1, 3 and 6 months after start of treatment and 1 week after end of tretment

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Golmand, MD, Study Director — AstraZeneca; Catherine Bonuccelli, Study Chair — AstraZeneca

REFERENCES:
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162
- [Derived] O'Connor RD, Patrick DL, Parasuraman B, Martin P, Goldman M. Comparison of patient-reported outcomes during treatment with adjustable- and fixed-dose budesonide/formoterol pressurized metered-dose inhaler versus fixed-dose fluticasone propionate/salmeterol dry powder inhaler in patients with asthma. J Asthma. 2010 Mar;47(2):217-23. doi: 10.3109/02770900903497154. PMID 20170333